CLINICAL TRIAL: NCT02660996
Title: Assessing the Effectiveness of the Advocate Lutheran General Survivorship Center Programs on Patients' Quality of Life, Distress Level, and Satisfaction
Brief Title: Effectiveness of the Advocate Lutheran General Survivorship Center Programs
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 5857
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2019-07

CONDITIONS: Cancer; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this observational study is to assess the effectiveness of the Advocate Lutheran General Survivorship Center's Programs by measuring the following outcomes of interest on participating patients:

1. Quality of life
2. Distress level
3. Satisfaction with the Survivorship Program

General Hypothesis: Patients who participate in at least four classes in a two month period will have higher scores on the post-class satisfaction, quality of life, and distress surveys compared to their pre-class surveys.

DETAILED DESCRIPTION:
* If a patient agrees to participate, written consent will be obtained by the study coordinators. Before the start of the first class at the Survivorship Center and after the patients have signed the consent and HIPAA authorization forms, patients will fill out three questionnaires. These include the standardized RAND 36 Health Survey, the Distress Thermometer, and a pilot survey regarding expectations and satisfaction with the Survivorship Program.
* The RAND-36 survey is a form that includes 36 questions and asks how patients feel their illness has impacted them and their lifestyle with scoring as noted. Pre-coded numeric values are recoded per the scoring key. They are scored so that a high score means patient is in better health, 0 being the worst and 10 being the best. Scores represent the percentage of total possible score achieved. Items in the same scale are averaged together to create the 8 scale scores. Missing data is not taken into account. The RAND 36-Item Health Survey 1.0 has been validated in previous studies. According to the VanderZee's study (1996), it was shown that the "internal consistency of the instrument was high with high convergent validity."
* The Distress Thermometer (DT) tool asks patients 39 questions about practical, family, emotional, religious, and physical problems in a "yes" or "no" format. A "yes" will scored as 0 and a "no" will be scored as 1. Therefore, the lower the stress level, the higher the score. The scores will be added for a total score. If the patient does show a high level of distress with a score above 12 on the Distress Thermometer after the four classes at the Survivorship Center, we will refer the patient back to his or her physician for further guidance and possible counseling.
* The Expectation Survey consists of eight questions that ask patients about their expectations for what they want/hope to get out of the Survivorship Program. Patients will rank their answers from 1 - 5 based on how much they agree with the statement (1 being not at all, 5 being very much). The scores for each eight questions will then be averaged.
* The Satisfaction Survey is also an eight question form that is much like the Expectation Survey. Patients will also indicate how satisfied with they are with the classes/courses at the Survivorship Center. The same scaling as above (1-5; 1 being not all agreeing with the statement and 5 being very much) with be used. These two surveys will be pilot tested for content relevance and readability level with current patients. Editions will be made as necessary. There will also be an open ended question at the end to ask patients what they would add to the classes to make them more beneficial.
* Participants will be asked to complete the Rand-36 SF, Distress Thermometer, and Satisfaction Survey after attending at least four Survivorship classes in a two month period.

ELIGIBILITY:
* Inclusion Criteria

  * Patients older than 18 years of age, any gender, and any race
  * Newly diagnosed with any type of cancer and now seeing one of the oncologists at the Advocate Lutheran General Hospital's Center for Advanced Care
  * Patients new to the Survivorship Center or only visited once
  * Must attend at least four classes in a two month period (any class, any time, any day)
  * Able to consent
  * English speaking patient
* Exclusion Criteria

  * Not a newly diagnosed cancer patient
  * Patients under the age of 18
  * Pregnant patients
  * Prisoners
  * Unable to consent
  * Non - English speaking patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed cancer patients who see one of the oncologists at The Advocate Lutheran General Hospital Center of for Advanced Care. Patients who older than 18 years of age, male or female, and any race are eligible. Patients who are new to the Survivorship Center or only visited once are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Quality of life | 6-8 months
  Questionnaire that includes 36 questions and asks how patients feel their illness has impacted them and their lifestyle with scoring as noted.

SECONDARY OUTCOMES:
Distress level | 6-8 months
  The tool asks patients 39 questions about practical, family, emotional, religious, and physical problems in a "yes" or "no" format. A "yes" will scored as 0 and a "no" will be scored as 1. Therefore, the lower the stress level, the higher the score. The scores will be added for a total score.
Satisfaction with the Survivorship Program | 6-8 months
  Questionnaire that includes 8 questions that indicate how satisfied the patients are with the classes offered at the Survivorship Center.

CONTACTS AND LOCATIONS:
Overall Officials: Sigrun Hallmeyer, MD, Principal Investigator — Advocate Lutheran General Hospital
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Conference presentation and publication